CLINICAL TRIAL: NCT06947954
Title: Nourish Intervention Trial
Brief Title: Nourish Clinical Trial
Acronym: Nourish_CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY20250330; CA2115405 (Other Grant/Funding Number: National Science Foundation)
Record Dates: First submitted 2025-04-25; First posted 2025-04-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Nutrition; Healthy
Keywords: Food literacy; Cooking skills
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nourish intervention then no intervention (Experimental): Subjects first participate in 9 weeks of weekly cooking classes, then no intervention for 9 weeks.
  Interventions: Behavioral: Nourish intervention then no intervention
- no intervention then nourish intervention (Experimental): Subjects receive no intervention for 9 weeks, then participate in 9 weeks of weekly cooking classes.
  Interventions: Behavioral: no intervention then Nourish intervention

INTERVENTIONS:
Behavioral: Nourish intervention then no intervention — Participants will attend a weekly in-person class with brief instructional video clips, hands-on cooking and tasting experiences. Participants will work individually and as part of small groups during instructional sessions. At the end of each class, participants will receive a grocery bundle and a kitchen gadget that serves both as an incentive and implementation support to promote improved cooking frequency and confidence. Participants will be asked to post photos of what they made with their groceries to an instant messaging software (GroupMe application) and be encouraged to engage with fellow classmates on GroupMe to encourage social support of cooking. After 9 weeks, participants crossover into the No Intervention group.
  Other Names: Intervention
  Arms: Nourish intervention then no intervention
Behavioral: no intervention then Nourish intervention — Participants will receive no intervention for 9 weeks. After 9 weeks, they crossover into the Nourish Intervention group where they will attend a weekly in-person class with brief instructional video clips, hands-on cooking and tasting experiences. Participants will work individually and as part of small groups during instructional sessions. At the end of each class, participants will receive a grocery bundle and a kitchen gadget that serves both as an incentive and implementation support to promote improved cooking frequency and confidence. Participants will be asked to post photos of what they made with their groceries to an instant messaging software (GroupMe application) and be encouraged to engage with fellow classmates on GroupMe to encourage social support of cooking.
  Other Names: Control
  Arms: no intervention then nourish intervention

SUMMARY:
The purpose of the research study is to learn more about the best ways to teach cooking and food skills to adults, and how cooking classes may help reduce one's stress and food waste, as well as improve their diet.

DETAILED DESCRIPTION:
Currently, 12.8% of Americans experience food insecurity, and food insecurity is associated with elevated perceived stress. Food literacy is proficiency in food-related skills and knowledge, including food preparation and cooking skills, basic nutrition knowledge, and the ability to prevent food waste. Recent research conducted in Australia suggests that food literacy interventions are associated with improved food security. Traditionally food literacy interventions take a recipe-based approach to culinary nutrition and lack information about key components of food literacy, such as food storage and food waste reduction techniques. However, recent research by the PI contends that recipes may be difficult for food insecure individuals to implement at home, given the challenge of procuring ingredients, suggesting the need for a new approach. In addition, food insecure households face additional environmental challenges, such as owning fewer cooking utensils, compared to food secure households. Based on the Social Cognitive Theory, the Nourish intervention addresses these limitations by incorporating food waste reduction, food storage knowledge, and improvisational cooking skills (cooking with what you have on hand) into food literacy and culinary nutrition education, as well as providing key cooking utensils. Eventually, the study team plans to test the impact of the Nourish intervention on food literacy, perceived stress, diet quality and food security to determine if food literacy interventions can positively impact perceived stress, diet, and food security. The present clinical trial will test the effectiveness of the Nourish intervention on household food waste, diet quality, and food and cooking skills and behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Ability to attend classes in person

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Food Waste Volume | Change from Baseline to 10 weeks post-randomization
  Food waste volume will be measured in grams using a study-provided food scale and waste log. Participants are asked to weigh discarded food and log the weight in a food waste tracking notebook for a period of 1 week prior to randomization at Baseline, and again for a period of 1 week at 10 weeks post-randomization. The outcome measure will use the difference in total volume of food waste between the two time points.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Prescott, PhD, Principal Investigator — Case Western Reserve University; Brenna Ellison, PhD, Principal Investigator — Purdue University
Locations (1):
- Community Recruitment, Cleveland, Ohio, United States